CLINICAL TRIAL: NCT06491147
Title: A Simple Model to Increase Residents' Confidence in Emergency Front of Neck Access (eFONA).
Brief Title: Increase Residents' Confidence in Emergency Front of Neck Access (eFONA).
Status: Not yet recruiting | Type: Observational
Sponsor: Kocaeli City Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2024-48
Record Dates: First submitted 2024-06-11; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Unexpected Difficult Airway

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- 1st year residency
  Interventions: Other: Emergency front of neck access
- 2nd year residency
  Interventions: Other: Emergency front of neck access
- 3rd year residency
  Interventions: Other: Emergency front of neck access
- 4th year residency
  Interventions: Other: Emergency front of neck access
- 5th year residency
  Interventions: Other: Emergency front of neck access

INTERVENTIONS:
Other: Emergency front of neck access — The algorithm in the DAS manual will be explained. Following this, the researcher will demonstrate the scalpel spark plug technique with a 4-step approach that is frequently used in skill teaching.
  In step 1 of this approach, the technique will be demonstrated without any verbal explanation.
  In the 2nd step, the technique will be demonstrated with verbal expression. In the 3rd step, the participant will be asked to have the trainer do it. In the 4th and last step, the participant will apply eFONA from start to finish.

SUMMARY:
Emergency front of neck access (eFONA) in a non-ventilated, non-oxygenated (CVCO) patient scenario is a life-saving and important competency for anesthesiologists to learn and even repeat intermittently. The Difficult Airway Society (DAS) guideline does not elaborate on how to conduct eFONA training, while the Canadian guideline states that successful performance of such rarely used skills requires regular practice in a simulation environment that focuses on technique and provides expert feedback. In this guideline, it was also mentioned that during training, procedures can be repeatedly performed in a simulate environment and interrupted for immediate feedback. In line with these recommendations, the investigators will create an easy, inexpensive, feasible and repeatable simulation-based learning environment in the operating room of the hospital. In this model study, it is aimed to teach the cricothyrotomy technique to anesthesiologists who have no experience in eFONA with an easy set up and to increase the confidence of the participants in this subject.

DETAILED DESCRIPTION:
Emergency front of neck access (eFONA) in a non-ventilated, non-oxygenated (CVCO) patient scenario is a life-saving and important competency for anesthesiologists to learn and even repeat intermittently. The Difficult Airway Society (DAS) guideline does not elaborate on how to conduct eFONA training, while the Canadian guideline states that successful performance of such rarely used skills requires regular practice in a simulation environment that focuses on technique and provides expert feedback. In this guideline, it was also mentioned that during training, procedures can be repeatedly performed in a simulate environment and interrupted for immediate feedback. In line with these recommendations, the investigators will create an easy, inexpensive, feasible and repeatable simulation-based learning environment in the operating room of the hospital. In this model study, it is aimed to teach the cricothyrotomy technique to anesthesiologists who have no experience in eFONA with an easy set up and to increase the confidence of the participants in this subject.

Participants will be divided into groups according to their duration of anesthesiology residency: 1st year, 2nd year, 3rd year, 4th and 5th year residents. A simple surgical airway delivery model will be created from the unused anesthesia circuit. The model will be described to the participants and anatomical markers will be explained: hyoid bone, thyroid cartilage, cricoid cartilage, cricothyroid membrane, tracheal rings. Then the algorithm in the DAS guidelines will be explained. Following this, the researcher will demonstrate the scalpel spark plug technique with a 4-step approach that is frequently used in skill teaching (4).

In step 1 of this approach, the technique will be demonstrated without any verbal explanation.

In the 2nd step, the technique will be demonstrated with verbal expression. In the 3rd step, the participant will be asked to have the trainer do it. In the 4th and last step, the participant will apply eFONA from start to finish.

Participants will apply all the steps on the model until they feel competent, then when the participants are ready, they will be asked to perform the technique by keeping a stopwatch. The stopwatch will be started when the participant takes the scalpel in his/her hand.

The circuit will be terminated when the balloon is inflated. In this way, a competitive learning environment will be created among the participants. Recorded values will be compared and minimum and maximum values will be determined. The participants will be asked the question "If you had to create an emergency FONA procedure, how long would it take you to open it?", the answers will be recorded and compared with the values after the research. Thus, it is aimed to increase the self-confidence of residents in eFONA.

ELIGIBILITY:
Inclusion Criteria:

* Working as an assistant doctor in Kocaeli City Hospital Anesthesiology and Reanimation Clinic

Exclusion Criteria:

* Those who have previously received training on FONA

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: After obtaining participant consent, anesthesiology residents with no previous emergency FONA experience will be included in the study. Participants who do not give consent and have previous experience will be excluded from the study. Participants will be divided into groups according to their duration of anesthesiology residency: 1st year, 2nd year, 3rd year, 4th and 5th year residents.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-06-30 (Estimated); Primary Completion 2024-12-21 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Emergency front of neck access training practice on a model | 6 months
  In this model study, it was aimed to teach the cricothyrotomy technique to anesthesiologists who had no experience in Emergency front of neck access (eFONA) and to increase the confidence of the participants in this subject. The participants who participated in the research will be asked the question "If you need to create an emergency FONA procedure, how long would you open it?", the answers will be recorded and compared with the values after the research. Thus, it is aimed to increase the self-confidence of residents in eFONA.

CONTACTS AND LOCATIONS:
Overall Officials: mehmet yilmaz, Principal Investigator — Kocaeli City Hospital Anesthesiology and Reanimation

IPD SHARING:
Plan to Share IPD: No